CLINICAL TRIAL: NCT00005590
Title: A Randomized, Prospective Double-Blind, Placebo-Controlled Trial of Prophylactic Oral Levofloxacin Following Chemotherapy for Lymphoma and Solid Tumors
Brief Title: Levofloxacin to Prevent Infection Following Chemotherapy in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRC-TU-SIGNIFICANT; CDR0000067666 (Registry Identifier: PDQ (Physician Data Query)); EU-99054
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2002-07

CONDITIONS: Brain and Central Nervous System Tumors; Breast Cancer; Extragonadal Germ Cell Tumor; Infection; Lung Cancer; Lymphoma; Ovarian Cancer; Small Intestine Cancer; Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent breast cancer; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; small intestine lymphoma; stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; unspecified adult solid tumor, protocol specific; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage II ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; extragonadal germ cell tumor; adult central nervous system germ cell tumor; primary central nervous system non-Hodgkin lymphoma; infection; intraocular lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage II small lymphocytic lymphoma; stage II marginal zone lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Breast Neoplasms; Infections; Lung Neoplasms; Lymphoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Small Cell Lung Carcinoma; Testicular Neoplasms; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
RATIONALE: Giving antibiotics may be effective in preventing or controlling early infection in patients receiving chemotherapy for solid tumors or lymphoma. It is not yet known if levofloxacin if effective in preventing infection.

PURPOSE: Randomized phase III trial to determine the effectiveness of levofloxacin in preventing infection in patients receiving chemotherapy for solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether prophylactic treatment with levofloxacin reduces the rate of clinical infection in patients receiving myelosuppressive antineoplastic chemotherapy for solid tumors or lymphoma.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to age (under 40 vs 40-59 vs 60 and over), type of cancer (non-Hodgkin's lymphoma vs Hodgkin's lymphoma vs breast vs germ cell vs small cell lung cancer vs other), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral levofloxacin once daily for 7 consecutive days during the expected neutrophil nadir of each chemotherapy course.
* Arm II: Patients receive an oral placebo once daily for 7 consecutive days as in arm I.

Treatment in both arms continues for up to 6 courses in the absence of unacceptable side effects or allergy or a clear continuing indication for the prophylactic use of antibacterial agents during subsequent courses.

PROJECTED ACCRUAL: A total of 1,500 patients (750 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of solid tumor, including but not limited to, the following:

  * Stage II-IV germ cell malignancy
  * Small cell lung cancer
  * Recurrent breast cancer OR
* Diagnosis of lymphoma
* About to start a program of antineoplastic chemotherapy for malignant disease that will regularly induce myelosuppression with a risk of temporary severe neutropenia (i.e., neutrophil count less than 500/mm3), but does not routinely require filgrastim (G-CSF) or stem cell support
* Not previously randomized into the Significant trial for a different multicourse chemotherapy program
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Creatinine normal OR
* Creatinine clearance greater than 40 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception in addition to oral contraceptive pills
* HIV negative
* No epilepsy
* No history of adverse events resulting from fluoroquinolone therapy (e.g., allergy or tendinitis)
* No concurrent use of a sunbed or exposure to strong sunlight

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent antibacterial therapy
* No other concurrent prophylactic antibacterial agents including cotrimoxazole prophylaxis against Pneumocystis carinii
* No iron supplements, sucralfate, or mineral antacids 2 hours before or after study medication
* Concurrent entry into other clinical trials allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08; Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Neil, MB, MA, BS, PhD, DTMH, MRCP, Study Chair — University Hospital Birmingham
Locations (1):
- University of Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Result] Cullen M, Steven N, Billingham L, Gaunt C, Hastings M, Simmonds P, Stuart N, Rea D, Bower M, Fernando I, Huddart R, Gollins S, Stanley A; Simple Investigation in Neutropenic Individuals of the Frequency of Infection after Chemotherapy +/- Antibiotic in a Number of Tumours (SIGNIFICANT) Trial Group. Antibacterial prophylaxis after chemotherapy for solid tumors and lymphomas. N Engl J Med. 2005 Sep 8;353(10):988-98. doi: 10.1056/NEJMoa050078. PMID 16148284